CLINICAL TRIAL: NCT03569605
Title: Promoting Physical Activity in Young Adult Cancer Survivors Using mHealth and Adaptive Tailored Feedback Strategies
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: University of South Carolina (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LCCC1707; R01CA204965 (NIH)
Record Dates: First submitted 2018-05-21; First posted 2018-06-26 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Physical Activity; Neoplasms; Neoplasms by Site; Cancer
Keywords: young adult; cancer survivor
MeSH Terms: conditions — Motor Activity; Neoplasms; Neoplasms by Site | interventions — Methods

STUDY DESIGN:
Intervention Model Description: After completing informed consent, 7-day PA assessment, weight measurement, and baseline questionnaires, participants will be randomly assigned with equal probability to 1 of 2 treatment groups: 1) self-help or 2) intervention. Future treatment assignments will be concealed from study staff who are recruiting and enrolling participants.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help (Active Comparator): Participants will receive an individual session, Fitbit activity tracker, and access to a secret Facebook group.
  Interventions: Behavioral: Intervention
- Intervention (Experimental): Participants will receive an individual session, Fitbit activity tracker, and access to a secret Facebook group, behavioral lessons, adaptive physical activity goals, tailored feedback summaries, and text messages.
  Interventions: Behavioral: Self-help

INTERVENTIONS:
Behavioral: Self-help — Participants will receive an individual session, Fitbit activity tracker, and access to a secret Facebook group.
  Other Names: Digital tools
  Arms: Intervention
Behavioral: Intervention — Participants will receive an individual session, Fitbit activity tracker, and access to a secret Facebook group with the addition of behavioral lessons, adaptive physical activity goals, tailored feedback summaries, and text messages.
  Other Names: Digital tools plus
  Arms: Self-help

SUMMARY:
To date, few interventions have been designed specifically to promote physical activity in young adult cancer survivors, nor used novel technologies for delivery; none have been successful in promoting long-term adherence to PA. The purpose of this randomized controlled trial is to test the efficacy of a theory-based, mobile physical activity intervention with adaptive goal-setting and tailored feedback that is aimed at increasing physical activity among young adult cancer survivors.

DETAILED DESCRIPTION:
There are over half a million young adult cancer survivors in the United States. Young adult cancer survivors are an underserved and vulnerable subgroup of survivors that experience increased risk over time for obesity and chronic diseases such as diabetes and cardiovascular disease. Increasing physical activity is a promising behavioral intervention that has positive effects on physical function, body composition, cardiovascular fitness, health-related quality of life, and depression, and may prevent cancer recurrence, new cancers and improve survival. To date, few interventions have been designed specifically to promote physical activity in young adult cancer survivors, nor used novel technologies for delivery; none have been successful in promoting long-term adherence to physical activity. This is a randomized controlled trial to test the efficacy of a theory-based, mobile physical activity intervention with adaptive goal-setting and tailored feedback that is aimed at increasing PA among young adult cancer survivors. Young adult cancer survivors (n=280), diagnosed between ages 18-39, will be recruited and randomized into one of two conditions: 1) activity tracker + Facebook group (Self-help) or 2) activity tracker + Facebook group + adaptive goal-setting and tailored feedback (Intervention). Young adult cancer survivors will receive a 6-month intervention followed by an additional 6 months of tapered contacts. Assessments of objectively-measured physical activity and other outcomes will be conducted at baseline, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently age 18-39
* Diagnosed with invasive malignancy between the ages of 18-39 years
* Diagnosed with invasive malignancy in the last 10 years with no evidence of progressive disease or second primary cancers
* Completed active cancer directed therapy (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention), except may be receiving "maintenance" therapy to prevent recurrences
* Have the ability to read, write and speak English
* No pre-existing medical condition(s) that preclude adherence to an unsupervised exercise program, including cardiovascular disease, congestive heart failure, pulmonary conditions, renal disease, and severe orthopedic conditions
* Not adhering to the American College of Sports Medicine recommendation of at least 150 moderate-to-vigorous physical activity minutes/week
* Have access to the Internet on at least a weekly basis
* Possession and usage of an Internet e-mail address or willingness to sign up for a free email account (e.g., gmail)
* Have mobile phone with text messaging plan
* Willing to be randomized to either arm
* Successful completion of accelerometer-assessed activity (i.e., at least 10 hours/day on 4 of 7 days) and return of the accelerometer in a pre-paid envelope at baseline

Exclusion Criteria:

* History of heart attack or stroke within past 6 months
* Untreated hypertension, hyperlipidemia, or diabetes, unless permission is provided by their health care provider
* Health problems which preclude ability to walk for physical activity
* Report a diagnosis of psychiatric diseases (schizophrenia, bipolar disorder, depression leading to hospitalization in the past year), drug or alcohol dependency.
* Report a past diagnosis of or treatment for a DSM-IV-TR eating disorder (anorexia nervosa or bulimia nervosa)
* Current participation in another physical activity or weight control program
* Currently using prescription weight loss medications
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Currently exercising > 150 minutes/week of moderate-to-vigorous intensity physical activity

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Minutes of total physical activity at 6 months: objective | Baseline, 6 months
  Change in objective levels of physical activity, as measured by accelerometry (ActiGraph), from baseline to 6 months. Participants will wear an accelerometer on their wrist during a 7 day period.

SECONDARY OUTCOMES:
Minutes of total physical activity at 6 months: self-report | Baseline, 6 months
  Change in self-report levels of physical activity, as measured by a modified version of the Godin Leisure Time Exercise Questionnaire, from baseline to 6 months. Participants report frequency of light, moderate and vigorous exercise, and average duration (minutes/week) for light, moderate and vigorous exercise bouts in a typical week. Scores for light, moderate and vigorous exercise are combined to compute total physical activity minutes/week.
Minutes of total physical activity at 12 months: objective | Baseline, 6 months, 12 months
  Change in levels of physical activity, as measured by accelerometry (ActiGraph), from baseline to 6 and 12 months. Participants will wear an accelerometer on their wrist during a 7 day period.
Minutes of total physical activity at 12 months: self-report | Baseline, 6 months, 12 months
  Change in levels of physical activity, as measured by a modified version of the Godin Leisure Time Exercise Questionnaire, from baseline to 6 and 12 months. Participants report frequency of light, moderate and vigorous exercise, and average duration (minutes) for light, moderate and vigorous exercise bouts in a typical week. Scores for light, moderate and vigorous exercise are combined to compute total physical activity minutes/week.
Minutes of light-intensity physical activity: objective | Baseline, 6 months, 12 months
  Change in levels of light-intensity physical activity, as measured by accelerometry (ActiGraph), from baseline to 6 and 12 months. Participants will wear an accelerometer on their wrist during a 7 day period.
Minutes of light-intensity physical activity: self-report | Baseline, 6 months, 12 months
  Change in levels of light-intensity physical activity, as measured by a modified version of the Godin Leisure Time Exercise Questionnaire, from baseline to 6 and 12 months. Participants report frequency of light, moderate and vigorous exercise, and average duration (minutes) for light, moderate and vigorous exercise bouts in a typical week. Scores for light-intensity physical activity are scored as minutes/week.
Minutes of moderate-to-vigorous intensity physical activity: objective | Baseline, 6 months, 12 months
  Change in levels of moderate-to-vigorous intensity physical activity, as measured by accelerometry (ActiGraph), from baseline to 6 and 12 months. Participants will wear an accelerometer on their wrist during a 7 day period.
Minutes of moderate-to-vigorous intensity physical activity: self-report | Baseline, 6 months, 12 months
  Change in levels of moderate-to-vigorous intensity physical activity, as measured by a modified version of the Godin Leisure Time Exercise Questionnaire, from baseline to 6 and 12 months. Participants report frequency of light, moderate and vigorous exercise, and average duration (minutes) for light, moderate and vigorous exercise bouts in a typical week. Scores for moderate and vigorous exercise are combined to compute moderate-to-vigorous intensity minutes/week.
Steps per day: objective | Baseline, 6 months, 12 months
  Change in steps per day, as measured by by accelerometry (ActiGraph), from baseline to 6 and 12 months. Participants will wear an accelerometer on their wrist during a 7 day period. Steps will be averaged over a minimum of 3 out of 7 days to calculate average daily step count.
Steps per day: Fitbit | Baseline, 6 months, 12 months
  Change in steps per day, as measured by by Fitbit, from baseline to 6 and 12 months. Participants will wear a Fitbit on their wrist during a 7 day period. Steps will be averaged over a minimum of 3 out of 7 days to calculate average daily step count.
Sedentary behavior | Baseline, 6 months, 12 months
  Change in sedentary behavior, as measured by self-report Sedentary Behavior Questionnaire, from baseline to 6 and 12 months. Participants will be asked to indicate the number of hours they spend on a typical weekday and typical weekend day doing a variety of sedentary activities. Responses range from 1 (none) to 9 (6 or more hours). To obtain weekly estimates of sedentary behavior, weekday hours are multiplied by 5 and weekend hours are multiplied by 2 and summed for total hours/week.
Weight | Baseline, 6 months, 12 months
  Change in weight, as measured objectively with digital scales, from baseline to 6 and 12 months.
Health-related quality of life: Medical Outcomes Study 36-Item Short Form (SF-36) | Baseline, 3 months, 6 months, 12 months
  Change in health-related quality of life, as measured using the Medical Outcomes Study 36-Item Short Form (SF-36), from baseline to 3, 6, and 12 months. The SF-36 asks respondents to rate their health and abilities to do their usual tasks. The SF-36 uses a variety of questions and response options and includes 8 subscales (physical functioning, role limitations due to physical health, role limitations due to emotional health, energy/fatigue, emotional well-being, social functioning, pain, and general health). Responses are coded on a scale of 0 to 100 where 0 is the worst possible health and 100 is the most favorable health score. The coded responses will be summed to yield a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score.
Health-related quality of life: Functional Assessment of Cancer Therapy-General (FACT-G) | Baseline, 3 months, 6 months, 12 months
  Change in health-related quality of life, as measured using the Functional Assessment of Cancer Therapy-General (FACT-G) survey, from baseline to 3, 6, and 12 months. The FACT-G is a 27-item measure specific to cancer patients to provide insight into cancer specific factors in four dimensions (physical, social/family, emotional, functional well-being). Participants will respond to a list of statements that tend to impact people with cancer by indicating how much they are impacted on a scale of 0 (not at all) to 4 (very much). Scores for negatively worded statements are reversed so that higher scores indicate positive health. Scores from the four dimensions can be summed to create a total score. Total possible scores range from 0 to 108, with higher scores indicating increased well being.
Behavioral capability | Baseline, 3 months, 6 months, 12 months
  Change in behavioral capability, as measured by self-report questionnaire, from baseline to 3, 6, and 12 months. Participants will be asked to rate how much they agree with six different statements. Responses range from 1 (strongly disagree) to 6 (strongly agree) and are averaged. Higher scores represent higher behavioral capability.
Self-efficacy for exercise | Baseline, 3 months, 6 months, 12 months
  Change in self-efficacy for exercise, as measured by the Self-Efficacy and Exercise Habits Survey, from baseline to 3, 6, and 12 months. Responses for two subscales (Sticking to it, Making time for exercise) are averaged to yield a score from 1 to 5, with higher values representing higher self-efficacy for exercise.
Self-regulation | Baseline, 3 months, 6 months, 12 months
  Change in self-regulation, as measured using by self-report questionnaire, from baseline to 3, 6, and 12 months. Responses to two subscales (Exercise goal-setting, Exercise planning and scheduling), ranging from 1 (does not describe) to 5 (describes completely), are averaged to yield two subscales. Higher subscale scores represent higher self-regulation.
Social support for exercise | Baseline, 3 months, 6 months, 12 months
  Change in social support for exercise, as measured by the Social Support for Exercise Survey, from baseline to 3, 6, and 12 months. Responses for three factors (Family participation, Friend participation, Friends on social networking sites participation), ranging from 1 to 5, are summed, with higher values representing higher social support for exercise.

OTHER OUTCOMES:
Mood | Baseline, 3 months, 6 months, 12 months
  Change in mood, as measured using the Profile of Mood States-Brief Form (POMS-BF), from baseline to 3, 6, and 12 months. The POMS-BF is a 30 item, self-report measure of six different mood states (such as "tense" or "angry") are rated based on how well each item describes the respondent's mood during the past week, including today. Items are rated on a 5-point scale with response options ranging from 0 (not at all) to 4 (extremely) with a global score range of 0 to 120 or individual domain scores on Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Lower scores indicate better mood state.
Depressive symptoms | Baseline, 3 months, 6 months, 12 months
  Change in depressive symptoms, as measured by the Center for Epidemiological Studies Depression Scale (CES-D), from baseline to 3, 6, and 12 months. The CES-D is a self-report depression scale including 20 items that relate to depressive feelings and behaviors during the past week. Response options range from 0 (rarely or none of the time) to 3 (most or almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Adherence to physical activity monitoring | Through study completion, 12 months
  Number of days physical activity tracked, as measured by Fitbit.
Adherence to self-weighing | Through study completion, 12 months
  Number of days weighed, as measured by digital scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carmina G. Valle, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Valle CG, Heiling HM, Deal AM, Diamond MA, Hales DP, Nezami BT, Rini CM, Pinto BM, LaRose JG, Tate DF. Examining sociodemographic and health-related characteristics as moderators of an mHealth intervention on physical activity outcomes in young adult cancer survivors. J Cancer Surviv. 2025 Oct;19(5):1611-1622. doi: 10.1007/s11764-024-01577-4. Epub 2024 Apr 12. PMID 38607515
- [Derived] Valle CG, Diamond MA, Heiling HM, Deal AM, Hales DP, Nezami BT, Pinto BM, LaRose JG, Rini CM, Tate DF. Effect of an mHealth intervention on physical activity outcomes among young adult cancer survivors: The IMPACT randomized controlled trial. Cancer. 2023 Feb 1;129(3):461-472. doi: 10.1002/cncr.34556. Epub 2022 Nov 29. PMID 36444676
- [Derived] Valle CG, Camp LN, Diamond M, Nezami BT, LaRose JG, Pinto BM, Tate DF. Recruitment of young adult cancer survivors into a randomized controlled trial of an mHealth physical activity intervention. Trials. 2022 Apr 4;23(1):254. doi: 10.1186/s13063-022-06148-5. PMID 35379294
- [Derived] Valle CG, Pinto BM, LaRose JG, Diamond M, Horrell LN, Nezami BT, Hatley KE, Coffman EM, Polzien K, Hales DP, Deal AM, Rini CM, Rosenstein DL, Tate DF. Promoting physical activity in young adult cancer survivors using mHealth and adaptive tailored feedback strategies: Design of the Improving Physical Activity after Cancer Treatment (IMPACT) randomized controlled trial. Contemp Clin Trials. 2021 Apr;103:106293. doi: 10.1016/j.cct.2021.106293. Epub 2021 Jan 27. PMID 33515784